CLINICAL TRIAL: NCT04048005
Title: RELATionship bEtween Lesion-level Invasive Fractional Flow Reserve AND Endothelial Wall Shear Stress the RELATE FFR and WSS Study
Brief Title: Relationship Between Fractional Flow Reserve/ Instantaneous Wave Free Ratio and Endothelial Wall Shear Stress
Acronym: RELATE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Collaborators: Politecnico di Torino (Unknown)
Responsible Party: Principal Investigator, Fabrizio D'Ascenzo, Medical Doctor, A.O.U. Città della Salute e della Scienza
Other Study IDs: RELATE FFR and WSS
Record Dates: First submitted 2019-08-04; First posted 2019-08-07 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Stable Angina; Acute Coronary Syndrome; Coronary Artery Disease
MeSH Terms: conditions — Angina, Stable; Acute Coronary Syndrome; Coronary Artery Disease | interventions — Fractional Flow Reserve, Myocardial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Fractional flow reserve
  Other Names: instantaneous wave free ratio

SUMMARY:
This study, designed as a retrospective registry, aims to investigate the relationship and potential interplay between fractional flow reserve (FFR) or instantaneous waves free ratio (iFR) with wall shear stress (WSS) in the context of intermediate coronary stenosis.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE Despite great advances in atherothrombosis science, the complex interplay of factors leading to plaque progression remains elusive. Specifically, the dynamics leading a stable plaque towards rupture and over imposed thrombosis are largely speculative. Wall shear stress (WSS), the mechanical force elicited by blood flow on the vessel walls, is emerging as a potent trigger of bio-humoral processes eventually leading to endothelial damage, plaque progression and destabilization.

Fractional flow reserve (FFR), assessing the aggregate hemodynamical significance of a stenosis on the subtended myocardium, stratifies the risk of major adverse cardiovascular events and reduces their occurrence when used to guide revascularization. While this event reduction is mainly driven by ischemia-caused urgent revascularization, it is emerging that FFR-guided revascularization may also reduce myocardial infarction.

While the physiological relationship between a lesion's FFR and resulting ischemia in the subtended myocardium is intuitive, the mechanisms linking FFR to atherothrombosis are less clearly defined.

Lesions with lower FFR are associated with adverse atherosclerotic plaque characteristics (APCs), however, the causative nexus of this relationship is not well established. It has been proposed both that the physiological base for this relation underlies in disturbed lesion hemodynamics, occurring at a greater extent as the degree of functional obstruction increases (i.e. FFR reduction drives APCs), and that APCs directly impair the vessel's vasodilatory reserve resulting in detrimental hyperemic perfusion (i.e. APCs drive FFR reduction).

WSS measures the regional tangential hemodynamic forces produced by viscous blood flow on the endothelium, which is established drivers of plaque progression and transformation toward an adverse plaque phenotype. Intriguingly, WSS may thus represent the missing link between FFR and atherothrombosis.

Few studies have focused on the interplay of FFR and WSS and the provided results are inconclusive (9, 10). This relation remains thus to be fully characterized.

This study will investigate the association of aggregate with regional hemodynamic forces as defined by the lesion-level relation of FFR or instantaneous wave-free ratio (iFR) and regional WSS across the lesion.

STUDY DESIGN This is a retrospective observational multi-center study, including consecutive patients who underwent coronary angiography at for symptom/ischemia-driven, suspected stable coronary artery disease or for acute coronary syndromes (ACS) with evidence of at least one lesion with 30-90% diameter-stenosis, that underwent subsequent iFR/FFR assessment.

Coronary angiography of the screened patients will be retrospectively evaluated by an experienced Interventional cardiologist and, if deemed suitable for baseline angiographic reconstruction will be included in this registry.

3-dimensional (3D) geometric reconstructions of each patient's target vessel will be created by using end-diastolic angiographic projections at least 25° apart. Computational fluid dynamics models will be applied to derive regional WSS values across the stenosis.

Clinical baseline characteristics and angiographic features obtained by visual and functional assessment, and 3-D reconstruction and computation, along with major adverse cardiovascular events, will be collected in a dedicated electronic form.

The analysts performing angiographic 3-D reconstruction and WSS computations will be blinded to FFR/iFR values and clinical data.

STUDY ENDPOINTS This study will investigate the association of aggregate and regional hemodynamic forces as established by the lesion-level relation of FFR/iFR with regional WSS across the lesion.

The association of regional WSS with major cardiovascular adverse events at available follow-up will be further evaluated to assess if lesion-level WSS might predict overall patient-level outcomes (in case of more than one lesion for a single patient, the lesion with the highest WSS will be considered for this analysis).

ELIGIBILITY:
Inclusion Criteria:

* Angiography performed for suspected symptom/ischemia-driven stable coronary artery disease or for acute coronary syndromes
* At least one lesion with 30-90% diameter stenosis at invasive angiography with FFR/iFR assessed (for patients with acute coronary syndromes, the invasive assessment will be performed on non-culprit stenosis
* Patient informed consent for data collection and publication in anonymous studies

Exclusion Criteria:

* Quality of angiographic frames not sufficient for 3D-reconstruction and/or computations
* Patients denying informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - The study will include any patient referred for coronary angiography at each involved center and with a subsequent invasive physiological assessment performed with FFR or iFR (or both) at operating physician's discretion on intermediate coronary stenosis (diameter of stenosis ranging from 30-90% at visual angiographic estimation).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Wall shear stress (WSS) / Fractional flow reserve (FFR) or instantaneous wave free ratio (iFR)correlation | WSS will be calculated after 3D coronary reconstruction, within one year after the completion of retrospective enrollement
  After 3-dimensional coronary reconstruction through dedicated software (Qangio XA 3D (MEDIS), WSS will be calculated through fluydodinamic equations across the entire coronary vessel and across coronary stenosis. WSS values predicting positive invasive FFR and iFR (according to their dichothomic established values of positivity, namely FFR < 0.8 and iFR < 0.89) measurements will be searched, along with any possible relationship between WSS and FFR/iFR as continuos values.
MACE (major adverse cardiovascular events) | MACE will be evaluated for each patients through study completion, an average of 1 year
  The association of regional WSS with major cardiovascular adverse events at available follow-up will be further evaluated to assess if lesion-level WSS might predict overall patient-level outcomes

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Ospedale di Rivoli, Rivoli
  - AOU Città della Salute e della Scienza di Torino, Torino
  - Ospedale San Giovanni Bosco, Torino

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ford TJ, Berry C, De Bruyne B, Yong ASC, Barlis P, Fearon WF, Ng MKC. Physiological Predictors of Acute Coronary Syndromes: Emerging Insights From the Plaque to the Vulnerable Patient. JACC Cardiovasc Interv. 2017 Dec 26;10(24):2539-2547. doi: 10.1016/j.jcin.2017.08.059. PMID 29268883
- [Background] Samady H, Eshtehardi P, McDaniel MC, Suo J, Dhawan SS, Maynard C, Timmins LH, Quyyumi AA, Giddens DP. Coronary artery wall shear stress is associated with progression and transformation of atherosclerotic plaque and arterial remodeling in patients with coronary artery disease. Circulation. 2011 Aug 16;124(7):779-88. doi: 10.1161/CIRCULATIONAHA.111.021824. Epub 2011 Jul 25. PMID 21788584
- [Background] Johnson NP, Toth GG, Lai D, Zhu H, Acar G, Agostoni P, Appelman Y, Arslan F, Barbato E, Chen SL, Di Serafino L, Dominguez-Franco AJ, Dupouy P, Esen AM, Esen OB, Hamilos M, Iwasaki K, Jensen LO, Jimenez-Navarro MF, Katritsis DG, Kocaman SA, Koo BK, Lopez-Palop R, Lorin JD, Miller LH, Muller O, Nam CW, Oud N, Puymirat E, Rieber J, Rioufol G, Rodes-Cabau J, Sedlis SP, Takeishi Y, Tonino PA, Van Belle E, Verna E, Werner GS, Fearon WF, Pijls NH, De Bruyne B, Gould KL. Prognostic value of fractional flow reserve: linking physiologic severity to clinical outcomes. J Am Coll Cardiol. 2014 Oct 21;64(16):1641-54. doi: 10.1016/j.jacc.2014.07.973. PMID 25323250
- [Background] De Bruyne B, Pijls NH, Kalesan B, Barbato E, Tonino PA, Piroth Z, Jagic N, Mobius-Winkler S, Rioufol G, Witt N, Kala P, MacCarthy P, Engstrom T, Oldroyd KG, Mavromatis K, Manoharan G, Verlee P, Frobert O, Curzen N, Johnson JB, Juni P, Fearon WF; FAME 2 Trial Investigators. Fractional flow reserve-guided PCI versus medical therapy in stable coronary disease. N Engl J Med. 2012 Sep 13;367(11):991-1001. doi: 10.1056/NEJMoa1205361. Epub 2012 Aug 27. PMID 22924638
- [Background] Zimmermann FM, Omerovic E, Fournier S, Kelbaek H, Johnson NP, Rothenbuhler M, Xaplanteris P, Abdel-Wahab M, Barbato E, Hofsten DE, Tonino PAL, Boxma-de Klerk BM, Fearon WF, Kober L, Smits PC, De Bruyne B, Pijls NHJ, Juni P, Engstrom T. Fractional flow reserve-guided percutaneous coronary intervention vs. medical therapy for patients with stable coronary lesions: meta-analysis of individual patient data. Eur Heart J. 2019 Jan 7;40(2):180-186. doi: 10.1093/eurheartj/ehy812. PMID 30596995
- [Background] Xaplanteris P, Fournier S, Pijls NHJ, Fearon WF, Barbato E, Tonino PAL, Engstrom T, Kaab S, Dambrink JH, Rioufol G, Toth GG, Piroth Z, Witt N, Frobert O, Kala P, Linke A, Jagic N, Mates M, Mavromatis K, Samady H, Irimpen A, Oldroyd K, Campo G, Rothenbuhler M, Juni P, De Bruyne B; FAME 2 Investigators. Five-Year Outcomes with PCI Guided by Fractional Flow Reserve. N Engl J Med. 2018 Jul 19;379(3):250-259. doi: 10.1056/NEJMoa1803538. Epub 2018 May 22. PMID 29785878
- [Background] Driessen RS, Stuijfzand WJ, Raijmakers PG, Danad I, Min JK, Leipsic JA, Ahmadi A, Narula J, van de Ven PM, Huisman MC, Lammertsma AA, van Rossum AC, van Royen N, Knaapen P. Effect of Plaque Burden and Morphology on Myocardial Blood Flow and Fractional Flow Reserve. J Am Coll Cardiol. 2018 Feb 6;71(5):499-509. doi: 10.1016/j.jacc.2017.11.054. PMID 29406855
- [Background] Kumar A, Thompson EW, Lefieux A, Molony DS, Davis EL, Chand N, Fournier S, Lee HS, Suh J, Sato K, Ko YA, Molloy D, Chandran K, Hosseini H, Gupta S, Milkas A, Gogas B, Chang HJ, Min JK, Fearon WF, Veneziani A, Giddens DP, King SB 3rd, De Bruyne B, Samady H. High Coronary Shear Stress in Patients With Coronary Artery Disease Predicts Myocardial Infarction. J Am Coll Cardiol. 2018 Oct 16;72(16):1926-1935. doi: 10.1016/j.jacc.2018.07.075. PMID 30309470
- [Background] Lee KE, Kim GT, Lee JS, Chung JH, Shin ES, Shim EB. A patient-specific virtual stenotic model of the coronary artery to analyze the relationship between fractional flow reserve and wall shear stress. Int J Cardiol. 2016 Nov 1;222:799-805. doi: 10.1016/j.ijcard.2016.07.153. Epub 2016 Aug 3. PMID 27522378